CLINICAL TRIAL: NCT02238704
Title: A Cluster-randomized, Non-inferiority Open-label Trial of the Impact of Supplementation Regimen on Consumption of Prenatal Calcium and Iron/Folic Acid Supplements and Adherence to Related Recommendations
Brief Title: Cornell University-Micronutrient Initiative Calcium Supplementation Study
Acronym: MICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Kenya Ministry of Health (Other Government); University of Nairobi (Other); Micronutrient Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB #: 1205003071; P414/01/2013 (Other: Kenyatta National Hospital Ethics Review Committee)
Record Dates: First submitted 2014-09-05; First posted 2014-09-12 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Preeclampsia
Keywords: Adherence; Calcium supplementation; Prevention of preeclampsia; Adherence to calcium supplementation
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen A (Experimental): 500mg elemental calcium (as CaCO3) + 200 microgram Vit D per administration, administered 2 times a day, at least 2hours apart with one administration of 60mg elemental iron (as FeSO4) at any time of the day
  Interventions: Dietary Supplement: Regimen A calcium and iron/folic acid
- Regimen B (Active Comparator): 500mg elemental calcium (as CaCO3) + 200 microgram Vit D per administration, administered 3 times a day, at least 2hours apart with one administration of 60mg elemental iron (as FeSO4) at any time of the day
  Interventions: Dietary Supplement: Regimen B calcium and iron/folic acid

INTERVENTIONS:
Dietary Supplement: Regimen A calcium and iron/folic acid — Comparison of recommended administration schedule for calcium and iron/folic acid supplements in pregnant women
  Arms: Regimen A
Dietary Supplement: Regimen B calcium and iron/folic acid — Comparison of recommended administration schedule for calcium and iron/folic acid supplements in pregnant women
  Arms: Regimen B

SUMMARY:
The World Health Organization (WHO) now recommends prenatal calcium supplementation for prevention of preeclampsia in populations with inadequate dietary intake. This study seeks to compare the effect of two dosing strategies on the amount of supplement ingested by pregnant women and adherence to related recommendations.

DETAILED DESCRIPTION:
This study is a non-inferiority trial that compares the effect of a dosing strategy involving lower overall dose and fewer administrations per day to the current WHO recommendation. The comparator arm, Regimen B, prescribes 3 doses per day (consistent with current WHO standard) and was found to be burdensome in qualitative studies. The experimental arm, Regimen A, prescribes 2 doses per day and has been associated with greater satisfaction. On face value Regimen A should result in 33% less amount of supplement ingested than Regimen B. However, we hypothesize that the difference in amount ingested, when rolled out in routine practice will be MUCH LESS than that BECAUSE THE LOWER DOSE REGIMEN RESULTS IN HIGHER LEVELS OF ADHERENCE. We hypothesize that THE DIFFERENCE IN AMOUNT CONSUMED WILL BE NEGLIGIBLE OR will not exceed 15%. Hence, we hypothesize that Regimen A is not inferior to Regimen B in terms of total amount of supplement ingested (within a 15% margin of inferiority).

ELIGIBILITY:
Inclusion Criteria:

* Attendance at ANC clinic in a primary care facility in Kakamega north

Exclusion Criteria:

* Gestational age < 16 weeks,
* Gestational age > 30 weeks,
* Dietary or medicinal consumption of adequate calcium (according to the screening survey),
* Intention to leave study community before 8weeks from date of interview

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1032 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Amount of calcium supplement ingested | 8 weeks after ANC consultation, during which recruitment into the study occurred
  This is the actual number of supplements ingested expressed as a percentage of the number of supplements expected to be ingested since the ANC consultation if 100% adherent to the current WHO recommendation.
  [Total number of calcium supplements consumed/(Number of days since last ANC consultation X 3)] X 100

SECONDARY OUTCOMES:
Adherence to related recommendations | 8 weeks after ANC consultation, during which recruitment into the study occurred
  Adherence to other features of the WHO recommendation (taking supplements with food).
Motivation | 8 weeks after ANC consultation, during which recruitment into the study occurred
  Motivation scores extracted from the survey instrument administered at follow up.
Self-efficacy | 8 weeks after ANC consultation, during which recruitment into the study occurred
  Self-efficacy scores extracted from the survey instrument administered at follow up.
Satisfaction | 8 weeks after ANC consultation, during which recruitment into the study occurred
  Satisfaction scores extracted from the survey instrument administered at follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Dickin, PhD, Principal Investigator — Cornell University
Locations (16):
- Kenya (16):
  - Chebwayi Health centre, Kakamega
  - Chegulo Health centre, Kakamega
  - Chevoso Health centre, Kakamega
  - Chimoi dispensary, Kakamega
  - Chombeli Health centre, Kakamega
  - Imbiakhalo Health centre, Kakamega
  - Kimangeti Health centre, Kakamega
  - Kuvasali Health centre, Kakamega
  - Malava district hospital, Kakamega
  - Manda Health centre, Kakamega
  - Miting'ongo Health centre, Kakamega
  - Mugai Health centre, Kakamega
  - Namagara Health centre, Kakamega
  - Shamberere Health centre, Kakamega
  - Shihome Health centre, Kakamega
  - Shivanga Health centre, Kakamega

REFERENCES:
- [Derived] Martin SL, Wawire V, Ombunda H, Li T, Sklar K, Tzehaie H, Wong A, Pelto GH, Omotayo MO, Chapleau GM, Stoltzfus RJ, Dickin KL. Integrating Calcium Supplementation into Facility-Based Antenatal Care Services in Western Kenya: A Qualitative Process Evaluation to Identify Implementation Barriers and Facilitators. Curr Dev Nutr. 2018 Aug 23;2(11):nzy068. doi: 10.1093/cdn/nzy068. eCollection 2018 Nov. PMID 30402593
- [Derived] Omotayo MO, Dickin KL, Pelletier DL, Mwanga EO, Kung'u JK, Stoltzfus RJ. A Simplified Regimen Compared with WHO Guidelines Decreases Antenatal Calcium Supplement Intake for Prevention of Preeclampsia in a Cluster-Randomized Noninferiority Trial in Rural Kenya. J Nutr. 2017 Oct;147(10):1986-1991. doi: 10.3945/jn.117.251926. Epub 2017 Sep 6. PMID 28878035
- [Derived] Martin SL, Omotayo MO, Pelto GH, Chapleau GM, Stoltzfus RJ, Dickin KL. Adherence-Specific Social Support Enhances Adherence to Calcium Supplementation Regimens among Pregnant Women. J Nutr. 2017 Apr;147(4):688-696. doi: 10.3945/jn.116.242503. Epub 2017 Mar 1. PMID 28250195